CLINICAL TRIAL: NCT04942704
Title: Development of Protocols and Methods for Image Processing and Enhancement of Magnetic Resonance Imaging (MRI) Data.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medic Vision Imaging Solutions Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: iQMR_CSP_01-00
Record Dates: First submitted 2021-06-21; First posted 2021-06-28 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: MRI Image Enhancement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non interventional Imaging - MRI — MRI Scanning using short protocols

SUMMARY:
The purpose of the study is to develop new methods for image processing and enhancement of MRI data. Different setting of acquisition parameters used in conventional clinical MRI protocols will be defined, to create "New Protocols".

The specific aim of this study is to assess and to improve the performance of our image processing methods, by comparing diagnostic qualities of images obtained by conventional MRI protocols with those obtained by corresponding New Protocols' and processed by our image enhancement method.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers for clinical MRI examination
* Patients undergoing clinical MRI examination
* Capable to provide an informed written consent form

Exclusion Criteria:

* Any contraindication to MRI scanning, such as pacemakers or heart rhythm disturbances, permanent cosmetics or certain metallic implants in the body (excluding dental implants).
* Age <18 years old
* Pregnancy
* Claustrophobia
* Decisional incapacity, mentally disabled,
* MRI exam under sedation or monitoring equipment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Total number of subjects expected to participate in this study is up to 100. The study population consists of patients who will go through their standard care MRI exam. Children, pregnant women and prisoners that are considered vulnerable population by federal regulation will not be included in this study. In addition, decisional incapacity subject will be excluded.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Image Signal to Noise Ratio (SNR) | Through study completion, an average of 2 months.
  Comparing the SNR of images obtained by conventional protocols with the corresponding New Protocols' processed images. The comparison will be performed by neuroradiologists, using a 7-point Likert-scale. Where higher the score, better the outcome (1 means unacceptable and 7 means excellent).
Image Resolution | Through study completion, an average of 2 months.
  Comparing the resolution of images obtained by conventional protocols with the corresponding New Protocols' processed images. The comparison will be performed by neuroradiologists, using a 7-point Likert-scale. Where higher the score, better the outcome (1 means unacceptable and 7 means excellent).
MRI contrast | Through study completion, an average of 2 months.
  Comparing MR contrast of images obtained by conventional protocols with the corresponding New Protocols' processed images. The comparison will be performed by neuroradiologists, using a 7-point Likert-scale. Where higher the score, better the outcome (1 means unacceptable and 7 means excellent).
Artifacts | Through study completion, an average of 2 months.
  Comparing artifacts of images obtained by conventional protocols with the corresponding New Protocols' processed images. The comparison will be performed by neuroradiologists, using a 7-point Likert-scale. Where higher the score, better the outcome (1 means unacceptable and 7 means excellent).
Diagnostic quality | Through study completion, an average of 2 months.
  Comparing diagnostic quality of images obtained by conventional protocols with the corresponding New Protocols' processed images. The comparison will be performed by neuroradiologists, using a 7-point Likert-scale. Where higher the score, better the outcome (1 means unacceptable and 7 means excellent).

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Medical Imaging, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No